CLINICAL TRIAL: NCT04235647
Title: A Nurse Led Intervention to Promote Physical Activity in Sedentary Older Adults With Cardio-vascular Risk Factors in the Outpatient Setting - a Randomized Controlled Trial
Brief Title: A Nurse Led Intervention to Promote Physical Activity
Acronym: STEP-IT-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DM-72
Record Dates: First submitted 2020-01-10; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Sedentary Behavior; Cardiovascular Risk Factor
Keywords: sedentary; older adults; risk factor; intervention; pedometer; clinical trial
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Older, sedentary adults (age 50-75 years) with and least one other cardiovascular risk-factor
  Interventions: Other: Nurse led tutorial on lifestyle management and pedometer hand-out; Other: Steps goal setting and supporting phone calls
- Control group (Active Comparator): Older, sedentary adults (age 50-75 years) with and least one other cardiovascular risk-factor
  Interventions: Other: Nurse led tutorial on lifestyle management and pedometer hand-out

INTERVENTIONS:
Other: Nurse led tutorial on lifestyle management and pedometer hand-out — Individual 10-minute nurse-led tutorial with distributed handouts on the health benefits of regular physical activity and pedometer hand-out
Other: Steps goal setting and supporting phone calls — A goal of minimum 7000 steps per day, phone calls to assess the goal meeting and to support goal achievement every 2 weeks
  Arms: Study group

SUMMARY:
Regular physical activity should be the essence of treatment in patients with cardiovascular risk factors. Unfortunately, these interventions are usually insufficiently promoted and therefore have only limited efficacy. The aim of the study was to determine the benefits of nurse led intervention to promote physical activity in sedentary older adults with cardio-vascular risk factors in the outpatient setting. Eligible patients are randomized in a 1:1 fashion to receive nurse led tutorial on life-style modification including pedometer hand-out with a daily goal of at least 7000 steps and supporting phone calls (study group) or without a goal or calls (control group). The primary end-point of the study is change in body weight. Secondary end-points include changes in resting heart rate, systolic and diastolic blood pressure, total cholesterol and fasting glucose and clinical outcomes at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* sedentary lifestyle defined as mean walking distance per day of no more than 3 km as reported by the patients;
* history of at least one of the following conditions: obesity (defined as body mass index ≥30 for I st degree obesity, ≥35 for second degree obesity and ≥40 for third degree obesity), hypertension, diabetes mellitus, dyslipidemia, stable coronary artery disease with or without prior myocardial infarction, peripheral arterial disease, stable arrhythmias, heart failure and/or prior stroke.

Exclusion Criteria:

* unstable clinical condition (in the form of unstable coronary artery disease or peripheral arterial disease, unstable heart failure or unstable arrhythmias);
* inability to undertake physical activity due to orthopedic reasons or other disabilities;
* planned changes in pharmacological treatment during the study period;
* lack of will to participate in the study and to sign the the written informed consent for the participation in the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Change in total body weight | 3 months

SECONDARY OUTCOMES:
Change in body mass index (BMI) | 3 months
Change in waist circumference | 3 months
Change in resting heart rate | 3 months
Change in resting blood pressure | 3 months
Change in total cholesterol concentration at fasting | 3 months
Change in glucose concentration at fasting | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz A. Małek, MD, PhD, Study Chair — Institute of Cardiology in Warsaw
Locations (1):
- NZOZ Arnika, Stare Babice, Ul. Rynek 10, Poland